CLINICAL TRIAL: NCT02810678
Title: Enhancing the Public Health Impact of Latent Tuberculosis (TB) Infection Diagnosis and Treatment: A Pragmatic Cluster Randomized Trial
Brief Title: Enhancing the Public Health Impact of Latent Tuberculosis (TB) Infection Diagnosis and Treatment
Acronym: ACT4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Dick Menzies, Director of Respiratory Epidemiology and Clinical Research Unit (RECRU), McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FND-143350
Record Dates: First submitted 2016-05-11; First posted 2016-06-23 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Latent Tuberculosis Infection
Keywords: Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No Intervention: Program runs as per usual. Minimal interference and visits from study staff. Main study outcomes evaluated in first and last 6 months of trial. Minimal visits to collect information on costing at control sites.
- Intervention (Active Comparator): Latent Tuberculosis Infection program evaluation & diagnosis: In intervention health facilities the current Latent Tuberculosis Infection program will be evaluated and gaps in the Latent Tuberculosis Infection cascade of care will be identified. Gaps in the current cascade will be quantified and solution proposed that are unique to the problems identified in each site. In phase 2 of the study low cost solutions will be implemented and the Latent Tuberculosis Infection program scaled up and improved. Study outcomes are evaluated in the first and last 6 months of trial. Costing evaluations are done throughout the trial.
  Interventions: Other: Latent Tuberculosis Infection program evaluation & diagnosis

INTERVENTIONS:
Other: Latent Tuberculosis Infection program evaluation & diagnosis
  Arms: Intervention

SUMMARY:
The study is a pragmatic cluster randomized trial that is being conducted in 5 countries, with sites in 4 cities in Canada, Benin, Ghana, Indonesia and Vietnam. The unit of randomization is the health facility (24 health facilities randomized). The trial tests a complex intervention-a two phase programmatic public health package which includes a standardized public health evaluation and analysis, to identify problems and barriers limiting Latent Tuberculosis Infection diagnosis and treatment among close contacts of active Tuberculosis cases. This will be followed by implementation of appropriate solutions and strengthening of the LTBI clinical program. The primary objective will be to estimate the increase the number of household contacts initiating LTBI treatment per newly diagnosed index patient, within 3 months of diagnosis of the index patient. A secondary objective is to evaluate the cost effectiveness of this two phase intervention. If successful, this approach can be expanded throughout these countries. After initial preparations, including administrative and ethical review, all participating sites will be randomized to intervention or control. Immediately after this, Phase 1 will begin in intervention sites with the standardized public health evaluation to identify barriers to LTBI diagnosis and treatment initiation and the selection of solutions to be used in Phase 2. To ensure standardization of data gathering research staff will use (i) current indicators of the Latent Tuberculosis Infection cascade of care in intervention facilities (number of contacts per index case registered, investigated, started on treatment and completing treatment) and (ii) interviewer administered questionnaires for patients with active pulmonary Tuberculosis, adult and child household contacts and clinic staff. These questionnaires will assess latent Tuberculosis-related knowledge, attitudes and beliefs from the perspective of these different participants. Results from intervention sites in Phase 1 will be analyzed, and used by the investigators, together with local public health officials, to decide on appropriate corrective solutions in each sites. Contact Investigation registries will also be developed with research staff from sites. In Phase 2, solutions for problems identified will be selected and implemented at the intervention sites, Contact Investigation registries will be implemented and clinical training will be provided to strengthen LTBI health care worker knowledge and clinical programs. Study outcomes and costs will be measured at all intervention and control sites throughout Phase 1 & 2. The main study will run for 18 months. Upon completion of the main study, a 1 year cross over study will be conducted where control sites will receive a streamlined version of the intervention and original intervention sites will be used to evaluate the sustainability of the intervention. Results will be disseminated within each country through existing links with National Tuberculosis Programs, and through international organizations such as the World Health Organization.

ELIGIBILITY:
Details vary depending on the study tool/measurement being taken. For Phase 1 questionniares (in 4 different populations) criteria are as follows:

1. Index case questionnaire:

   Inclusion Criteria:
   * Newly diagnosed patients with microbiologically confirmed active pulmonary Tuberculosis (Pulmonary Tuberculosis - smear or culture or GeneXpert positive or Nucleic Acid Amplification test (NAAT)
   * Age ≥ 18 years old
   * At least 1 Household contact, with contact investigation underway
   * Signed informed consent

   Exclusion Criteria:
   * Health care worker
   * Only extra-pulmonary Tuberculosis
2. Household contacts questionnaire

   Inclusion Criteria:
   * Age ≥ 18 years old
   * Informed consent signed
   * Sleeps in the same house at least 1 night per week during the past 3 months with person who has confirmed active Tuberculosis OR
   * Spent more than one hour per day in the house for at least 5 days per week with person who has active Tuberculosis - in the past 3 months

   Exclusion criteria:
   * Adult contact (age ≥ 18) who has already completed the child contact questionnaire
   * Currently has active Tuberculosis
   * Health Care worker
3. Health Care worker questionnaire:

   Inclusion criteria:
   * Health care worker involved in care of Tuberculosis patients, and/or their contacts
   * Age ≥ 18 years old
   * Signed informed consent

   Exclusion criteria:

   - Has ACTIVE TUBERCULOSIS (currently or in the past)
4. Parents of Children (under 5 years of age) who were Household contact

Inclusion criteria:

* Age ≥ 18 years old
* Signed informed consent
* Parent/legal guardian/responsible caregiver of child under 5 years of age

And one of the following two mandatory eligibility criteria:

* Child sleeps in the same house at least 1 night per week during the past 3 months with person who has active pulmonary Tuberculosis OR
* Child spent more than one hour per day in the house for at least 5 days per week with person who has active pulmonary Tuberculosis ( in the past 3 months)

Exclusion criteria:

* The parent is the source (Index) case
* The parents is an Aadult contact who has already completed the contact questionnaire for adults
* The child currently has active Tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in the number of household contacts (HHC) initiating treatment per newly diagnosed TB index patient within 3- 4 months from index patient diagnosis, between Phase 1 and Phase 2 | The primary outcome will be recorded at all health facilities for the full duration of phase 1 (6 months) and for the last 6 months of phase 2.
  A new TB index patient will be microbiologically confirmed using AFB smear, culture, and/or molecular tests such as Xpert®MTB/RIF, depending on local protocols. A HHC will be defined as someone who slept in the same house at least one night per week, or spent more than one hour in the house at least five days per week, on average, over the preceding 3 months. The house will be defined as the dwelling, or buildings, which the family unit occupies and uses regularly. In each of the 6 month periods, the total number of index patients, the number of their contacts who were recorded in clinic documents, and the number of these HHC who initiate LTBI therapy will be collected in both the control and intervention arms. For TB index patients diagnosed towards the end of each 6-month period in most sites we will allow up to 3 or 4 additional months for the HHC to be started on LTBI treatment.

SECONDARY OUTCOMES:
Health system costs related to the implementation of the LTBI program evaluation and strengthening approach | 18 months
  Throughout the trial, costs related to the implementation of the LTBI program evaluation and strengthening will be measured in each setting, using time and activity logs for research staff, investigators, health care workers and management staff involved in implementation. Country specific budgets will be used to obtain expenditures related to services, supplies and materials. To estimate LTBI related health system personnel costs, time and motion studies will be conducted at the start of phase 1 and the end of phase 2.
Cross-over | 12 months
  To evaluate the sustained effect of this complex intervention for one year after the end of the randomized trial - at original intervention sites.To evaluate the costs, and impact of a stream-lined Phase 1 and 2 - administered to control sites, after the 18 month trial.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, MD, Principal Investigator — Research Institute of McGill University Health Centre
Locations (8):
- Centre de Pneumo-Phthysiologie, Cotonou, Benin
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Montreal Chest Institute, Montreal, Quebec
- Komfo Anokye Teaching Hospital (KATH), Kumasi, Ghana
- University Padjadjaran (UNPAD), Bandung, Indonesia
- Vietnam national university, Hanoi, Vietnam

REFERENCES:
- [Derived] Menzies D, Obeng J, Hadisoemarto P, Ruslami R, Adjobimey M, Fisher D, Barss L, Bedingfield N, Long R, Paulsen C, Johnston J, Romanowski K, Cook VJ, Fox GJ, Nguyen TA, Valiquette C, Oxlade O, Fregonese F, Benedetti A. Sustainability and impact of an intervention to improve initiation of tuberculosis preventive treatment: results from a follow-up study of the ACT4 randomized trial. EClinicalMedicine. 2024 Mar 28;71:102546. doi: 10.1016/j.eclinm.2024.102546. eCollection 2024 May. PMID 38586588
- [Derived] Oxlade O, Benedetti A, Adjobimey M, Alsdurf H, Anagonou S, Cook VJ, Fisher D, Fox GJ, Fregonese F, Hadisoemarto P, Hill PC, Johnston J, Khan FA, Long R, Nguyen NV, Nguyen TA, Obeng J, Ruslami R, Schwartzman K, Trajman A, Valiquette C, Menzies D. Effectiveness and cost-effectiveness of a health systems intervention for latent tuberculosis infection management (ACT4): a cluster-randomised trial. Lancet Public Health. 2021 May;6(5):e272-e282. doi: 10.1016/S2468-2667(20)30261-9. Epub 2021 Mar 22. PMID 33765453
- [Derived] Oxlade O, Trajman A, Benedetti A, Adjobimey M, Cook VJ, Fisher D, Fox GJ, Fregonese F, Hadisoemarto P, Hill PC, Johnston J, Long R, Obeng J, Ruslami R, Valiquette C, Menzies D. Enhancing the public health impact of latent tuberculosis infection diagnosis and treatment (ACT4): protocol for a cluster randomised trial. BMJ Open. 2019 Mar 20;9(3):e025831. doi: 10.1136/bmjopen-2018-025831. PMID 30898826

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT02810678/SAP_000.pdf